CLINICAL TRIAL: NCT02361580
Title: Impact of Keeping a Personal Recovery Diary on Upper Extremity Disability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principal Investigator left the institution so the study was stopped before completing enrollment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Chief of Hand and Upper Extremity Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002781
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Acute Injury of Upper Extremity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diary (Experimental): Subjects that are randomized to the diary group will be told to keep a diary of their recovery. The study is focusing on the effect of keeping a diary on disability, rather than the content of the diary.
  Interventions: Other: Diary
- No Diary (No Intervention): Control Group

INTERVENTIONS:
Other: Diary — Subject keeps diary of recovery
  Arms: Diary

SUMMARY:
Primary null hypothesis:

• Keeping a personal diary has no effect on upper-extremity disability (assessed w/ PROMIS [Patient Reported Outcome Measurement Information System] upper extremity) 8 weeks after injury.

Secondary null hypotheses:

* Keeping a personal diary has no effect on avoidance of painful activities (assessed w/ PROMIS pain interference) 8 weeks after injury.
* Keeping a personal diary has no effect on symptoms of depression (assessed w/ PROMIS depression) 8 weeks after injury.
* There are no factors associated with upper-extremity disability 8 weeks after injury.

DETAILED DESCRIPTION:
Recovery from injury can be counterintuitive and taxing. It is natural to feel protective and prepare for the worst. Healthy exercises can seem unwise. It can seem like things are taking too long or getting off track. We have noticed that small improvements such as being able to resume a cherished activity (e.g. knitting or swimming) or achieving some success with exercises (e.g. obtaining full supination after fracture of the distal radius), can help patients feel like things are going to be okay. That feeling seems to make it easier to do exercises and resume function activities.

We wonder if awareness of this process (mindfulness) would help patients recover more rapidly. Keeping a journal is one method for encouraging mindfulness. It allows patients to express themselves and tell their stories. There is evidence that such "narrative medicine" can be healing. We anticipate that patients who perceive little or no progress will be able to look back on how they were feeling earlier on and appreciate that things are moving in the right direction. We also hope that their journal material might be useful for other patients that are having trouble seeing the "light at the end of the tunnel", so as part of this study, we will get permission to use their quotes anonymously in future patient care materials and future research. To our knowledge, research on the impact of keeping a personal diary/journal of recovery is scant, particularly pertaining to recovery from upper extremity trauma.

Explanatory variables:

* Diary or no Diary
* Diagnosis (fracture, sprain, contusion, skin laceration, complex laceration [tendon, nerve])
* Location (hand, wrist, forearm, elbow, arm, shoulder)
* Sex
* Age
* Education
* Work status
* Insurance (worker's compensation, private, public, other)
* Visit type
* Prior treatment received
* Other pain conditions
* Smoking status
* Marital status
* Physical or Occupational Therapy

ELIGIBILITY:
Inclusion Criteria:

* All new patients (>18 years) with an acute injury of the upper extremity (fracture, laceration, sprain, contusion)
* English fluency and literacy
* Able to take informed consent

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diary | No Diary
Started | 6 | 3
Completed | 0 | 0
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diary | No Diary | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (19) | 54 (10) | 52 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Disability Measured by PROMIS Upper Extremity
Description: Upper Extremity Disability measured by PROMIS Upper Extremity
Time Frame: 8 weeks
Population: All of the subjects were lost to follow up in both groups.
Arm/Group | Diary | No Diary
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Avoidance of Painful Activities Measured by PROMIS Pain Interference
Description: Avoidance of painful activities measured by PROMIS Pain Interference
Time Frame: 8 weeks
Population: All of the subjects were lost to follow up.
Arm/Group | Diary | No Diary
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Symptoms of Depression Measured by PROMIS Depression
Description: Symptoms of depression measured by PROMIS Depression
Time Frame: 8 weeks
Population: All of the subjects were lost to follow up.
Arm/Group | Diary | No Diary
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Diary | No Diary
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes